CLINICAL TRIAL: NCT02010138
Title: Extent of Internal Limiting Membrane Removal and Its Impact on Outcomes of Macular Hole Surgery
Brief Title: Extent of ILM Removal and Its Impact on Outcomes of MH Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-07-083
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Macular Holes
Keywords: Internal Limiting Membrane; Metamorphopsia
MeSH Terms: conditions — Retinal Perforations; Vision Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Small Extent Group (SG) (Active Comparator): Patients who were scheduled for surgery for idiopathic macular hole were randomly assigned to the SG. The small-extent peeling was performed in SG.
  Interventions: Procedure: small-extent peeling
- Large Extent Group (LG) (Active Comparator): Patients who were scheduled for surgery for idiopathic macular hole were randomly assigned to the LG. The large-extent peeling was performed in LG.
  Interventions: Procedure: large-extent peeling

INTERVENTIONS:
Procedure: small-extent peeling — The internal limiting membrane was peeled in round shape with the radius of 0.75-disc diameter radius (1.5-disc diameter in total) centering at the center of the macular hole.
  Arms: Small Extent Group (SG)
Procedure: large-extent peeling — The internal limiting membrane was peeled in round shape with the radius of 1.5-disc diameter radius (3.0-disc diameter in total) centering at the center of the macular hole.
  Arms: Large Extent Group (LG)

SUMMARY:
Eligible patients who were scheduled for surgery for idiopathic macular hole (MH) were equally randomized to small extent group or large extent group depending on the extent of internal limiting membrane (ILM) to be removed. The ILM was peeled in round shape with the radius of either 0.75-disc diameter or 1.5-disc diameter according to the group. The primary analysis was conducted to identify the difference of functional and anatomical outcomes between the two groups. Subsequent analysis was performed to reveal the relationship between the functional and anatomical outcomes.

DETAILED DESCRIPTION:
This randomized clinical trial was performed at a single center. Patients who were scheduled for surgery for idiopathic macular hole (MH) were enrolled. Eligible patients were equally randomized to small extent group or large extent group depending on the extent of ILM to be removed. Random numbers were generated through computerized block-randomization.

A standard 3-port pars plana vitrectomy was performed by a single surgeon using 23-gauge vitrectomy system, with a 1-step scleral tunnel incision. After posterior vitreous detachment was achieved, peeling of the ILM was performed by an end gripping forceps with the assistance of indocyanine green dye. The ILM was peeled in round shape with the radius of either 0.75-disc diameter or 1.5-disc diameter centering at the center of the MH according to the pre-assigned group. This was followed by a complete fluid-gas exchange, and all patients were encouraged to maintain a face-down position for at least 5 days postoperatively.

Postoperative measurements of BCVA and M-score were conducted at 2- and 6-month follow-up visits by independent masked observers. The first postoperative SD-OCT scanning was usually conducted at 1 to 2 weeks after operation according to the intraocular gas status. Then, OCT scans were conducted at follow-up visits 2, and 6 months postoperatively. The same experienced examiner conducted all the OCT scans on all subjects.

Comparison of anatomical closure, BCVA, M-score, Δ BCVA, and Δ M-score were primarily performed between the two groups. Then, the parameters measured from OCT scans with changes in ETDRS visual acuity and M-score were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic macular hole

Exclusion Criteria:

* macular hole associated with other causative diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Degree of foveal elongation | postoperative 6months

SECONDARY OUTCOMES:
metamorphopsia | 6months

OTHER OUTCOMES:
change in visual acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kunho Bae, MD, Principal Investigator — Department of Ophthalmology, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea